CLINICAL TRIAL: NCT05518188
Title: A Phase 1/2 Open-label Intrathecal Administration of MELPIDA to Determine Its Safety and Efficacy for Patients with Spastic Paraplegia Type 50 (SPG50) Caused by Mutation in the AP4M1 Gene.
Brief Title: Melpida: Recombinant Adeno-associated Virus (serotype 9) Encoding a Codon Optimized Human AP4M1 Transgene (hAP4M1opt)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elpida Therapeutics SPC (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND No 028202; Serial No 0000
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-11

CONDITIONS: Spasticity, Muscle; Microcephaly; Intellectual Deficiency; Growth Retardation; SPG50; Spastic Paraplegia
MeSH Terms: conditions — Muscle Spasticity; Microcephaly; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): MELPIDA, a gene therapy product
  Interventions: Biological: MELPIDA

INTERVENTIONS:
Biological: MELPIDA — MELPIDA, a recombinant serotype 9 adeno-associated virus (AAV) encoding a codon-optimized human AP4M1 transgene

SUMMARY:
MELPIDA is proposed for the treatment of subjects with SPG50 and targets neuronal cells to deliver a fully functional human AP4M1 cDNA copy via intrathecal injection to counter the associated neuronal loss. Outcomes will evaluate the safety and tolerability of a single dose of MELPIDA, which will be measured by the treatment-associated adverse events (AEs) and serious adverse events (SAEs). Secondarily, the trial will explore efficacy in terms of disease burden assessments.

DETAILED DESCRIPTION:
MELPIDA is a gene therapy product being developed for the treatment of Spastic Paraplegia Type 50 (SPG50), which is one of a group of four genetic disorders (SPG47, SPG50, SPG51 and SPG52) comprising AP-4 related Spastic Paraplegia (AP4-SPG). Inherited in an autosomal recessive pattern, AP-4- SPG is caused by biallelic pathogenic variants in one of 4 genes that encode components of the heterotrimeric adaptor protein complex 4 (AP4). Mutations in any of the components result in disrupted AP-4 function, and result in a common, shared clinical phenotype. Adaptor protein complexes such as AP-4 play key roles in signal-mediated trafficking of integral membrane proteins. They mediate vesicle formation and the cargo contained within these vesicles. While the precise function of the AP-4 complex is not fully understood, recent data suggests it plays an important role in protein sorting through the golgi, including regulation of trafficking of components required for autophagy. Deficiency in AP-4 leads to progressive neurodegeneration.

AP-4-HSP is an ultra-rare autosomal recessive disease with ~250 patients identified worldwide, 110 of which have the SPG50 subtype. There are approximately 21 patients with SPG50 in North America (OMIM #612936), ClinicalTrials.gov Identifier: NCT04712812. SPG50 is caused by biallelic pathogenic variants in the AP4M1 gene.

The AP4-deficiency syndrome (AP-4-HSP) is characterized by progressive spasticity, microcephaly, intellectual deficiency, dysmorphic traits, and growth retardation. Symptoms of AP-4-HSP begin in infancy, though patients are often not correctly identified and diagnosed until age 5 to 10 years. Patients experience progressive spastic paraplegia in the first decade of life, resulting in quadriplegia by adolescence or early adulthood with associated wheelchair dependence. There is also the presence of severe, progressive cognitive impairment. Epilepsy is an important co-morbidity present in the majority of cases. Only a few affected individuals have been identified to survive beyond age 30 year, though the extent of early mortality is yet to be fully elucidated.

Based on an AP-4-HSP natural history study currently in progress at Boston Children's Hospital (BCH), it is evident that disease severity ranges from child to child, but that most children fall into the severely affected (i.e. severe spasticity with paralysis and severe cognitive impairment) category. A small proportion of children, considered least severe, are able to speak in short sentences, walk with an abnormal gait, and have few to no seizures early on in the disease (less than 10 years of age). However, most children in this less severe category still experience progressive decline, ultimately losing the ability to walk and becoming quadriplegic between the ages of 10 and 20 years.

The majority of children with the SPG50 subtype of AP-4-HSP conform to a severe presentation, and are completely non-verbal, have microcephaly, never walk, have epilepsy and are severely cognitively impaired by the age of 10. It is not known how patients are affected later in life as very few have been identified beyond the age of 30. SPG50 is thus a degenerative neurological disease, affecting both cognitive and motor capabilities. Importantly, there is significant care giver burden, as all patients eventually require complete support for all activities of daily living from family and/or caregivers. There are no treatments currently available for patients with SPG50.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 months-10 years old
2. Confirmed diagnosis of SPG50 disease by:

   1. Genomic DNA mutation analysis demonstrating homozygous or compound heterozygous, confirmed pathogenic variants in the AP4M1 gene
   2. Clinical history or examination features consistent with SPG50 and that include neurologic dysfunction
3. Parent/legal guardian willing to provide written informed consent for their child prior to participation in the study
4. Subject able to comply with all protocol requirements and procedures
5. Ability to stand for more than 5 seconds OR
6. Ability to take 5 steps independently or with a walker OR
7. Modified Ashworth Scale score 2 or below (Ankles).

Exclusion Criteria:

1. Inability to participate in study procedures (as determined by the site investigator)
2. Presence of a concomitant medical condition that precludes lumbar puncture (LP) or use of anesthetics
3. History of bleeding disorder or any other medical condition or circumstance in which lumbar puncture is contraindicated according to local institutional policy
4. Inability to be safely sedated in the opinion of the clinical anesthesiologist
5. Active infection, at the time of dosing, based on clinical observations
6. Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer
7. Inability of the patient to undergo MRI according to local institutional policy
8. Inability of the patient to undergo any other procedure required in this study
9. The presence of significant non-SPG50 related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study
10. Have received an investigational drug within 30 days prior to screening or plan to receive an investigational drug (other than gene therapy) during the study.
11. Enrollment and participation in another interventional clinical trial
12. Contraindication to MELPIDA or any of its ingredients
13. Contraindication to any of the immune suppression medications used in this study
14. Clinically significant abnormal laboratory values (GGT, ALT, and AST, or total bilirubin > 3 × ULN, creatinine ≥ 1.5 mg/dL, hemoglobin [Hgb] < 6 or > 20 g/dL; white blood cell [WBC] > 20,000 per cmm) prior to gene replacement therapy.

Ages: 4 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of unanticipated treatment-related toxicities, Grade 3 or higher in participants with SPG50 | 60 months
  Incidence of unanticipated treatment-related toxicities, Grade 3 or higher, in participants with SPG50 will be determined from the collection of occurrence and severity of serious adverse events (SAEs). Adverse events will be determined according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Stability or improvement in spasticity in participants with SPG50 as measured by the Modified Ashworth scale (MAS) | 60 months
  Stability or improvement in spasticity in participants with SPG50 is measured by the Modified Ashworth scale (MAS) which is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion. Possible scores range from 0-4 where lower scores indicate better outcome.
Stability or improvement in spasticity in participants with SPG50 as measured by the Tardieu scale | 60 months
  Stability or improvement in spasticity in participants with SPG50 is measured by the Tardieu scale which quantifies muscle spasticity by assessing the response of the muscle to stretch applied at specified velocities. Possible scores range from 0-5 where lower scores indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susan T. Iannaccone, MD, FAAN, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Cure SPG50
Supporting Information: Study Protocol, SAP, ICF
Time Frame: End of study

REFERENCES:
- [Derived] Agianda HAP, Kim HM, Battaglia N, Rong J, Tam A, Gonzalez Saez-Diez E, Boerkoel CF, Saffari A, Quiroz V, Schierbaum L, Zaman Z, Bernardi K, Ebrahimi-Fakhari D. Diagnostic Utility of the ATG9A Ratio in AP-4-Associated Hereditary Spastic Paraplegia. Ann Clin Transl Neurol. 2026 Jan 5. doi: 10.1002/acn3.70308. Online ahead of print. PMID 41491634